CLINICAL TRIAL: NCT05885659
Title: A Multicomponent Smoking Cessation Program for Adults With Type 2 Diabetes Mellitus: A Study Protocol of a Randomized Controlled Trial (DiMe-SALUD2 Project)
Brief Title: Smoking Cessation Program for Adults With Type 2 Diabetes Mellitus (DiMe-SALUD2 Project)
Acronym: DiMe-SALUD2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Andalusian Plan for Research, Development, and Innovation (Unknown)
Responsible Party: Principal Investigator, Carla Lopez Nunez, Principal Investigator: Carla López-Núñez, Ph.D. Department of Personality, Assessment and Psychological Treatments, School of Psychology, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ProyExcel_00669
Record Dates: First submitted 2023-05-04; First posted 2023-06-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Tobacco Use Disorder; Diabetes Mellitus, Type 2
Keywords: Smoking cessation; Tobacco Use Disorder; Type 2 Diabetes Mellitus; Randomized controlled trial
MeSH Terms: conditions — Tobacco Use Disorder; Diabetes Mellitus, Type 2; Smoking Cessation | interventions — Control Groups; Waiting Lists

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of three groups (Control Group, Experimental Group 1, Experimental Group 2). A member of the research team who will not be directly involved in the trial (i.e., development of the assessments and treatment sessions) will create a simple computer-generated randomization sequence using Research Randomizer software (version 4.0, Urbaniak GC and Plous S, Middletown, CT, USA; http://www.randomizer.org).
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers who will develop the pre-treatment evaluation and the intervention program will not participate in the randomization process. The patients will be masked with respect to the study group to which they will belong. On the other hand, psychologists who develop the intervention must necessarily know the type of treatment they are applying (in trials where interventions of a psychological nature are assessed, it is usually not possible to mask the professionals implementing the intervention). However, such psychologists will not participate in the randomization process of the participants or in the analysis of the data, therefore the possible biases of the evaluator regarding such tasks will be deleted. Moreover, the following strategies will be carried out: 1) specialized training on the treatments to be applied, emphasizing the need to maintain masking of the participants; 2) professionals will rotate through all treatment modalities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (waiting list) (Other): T2DM in the control group will receive brief psychoeducation advice about smoking cessation as well as a general smoking cessation brochure/ booklet.
  Interventions: Other: Control group (waiting list)
- Experimental 1: Cognitive-behavioral treatment (CBT) for smoking cessation (Active Comparator): CBT for smoking cessation, implemented in group-based sessions over an eight-week period. Includes three different stages: (1) Motivational interviewing to stop smoking; (2) Smoking cessation, focused on nicotine fading from the first to the fourth session; (3) Maintenance of abstinence and relapse prevention strategies from the fifth session onwards.
  Interventions: Behavioral: Cognitive Behavioral Treatment (CBT) for smoking cessation
- Experimental 2: CBT for smoking cessation + DiMeSALUD2 protocol (Active Comparator): In this group, a training protocol on healthy lifestyle habits and self-management of T2DM will be carried out added to usual care (CBT for smoking cessation), including healthy lifestyle habits (dietary control and healthy nutrition, physical exercise, and glycemic control).
  Interventions: Behavioral: CBT for smoking cessation + DiMeSALUD2 protocol

INTERVENTIONS:
Other: Control group (waiting list) — T2DM in the control group will receive brief psychoeducation advice about smoking cessation as well as a general smoking cessation brochure/ booklet. Participants assigned to this control group will participate in the scheduled assessments (pre- and post-treatment, 1-month, 6-months and 12-months follow-ups) but without receiving any of the intensive treatments previously described (CBT vs. CBT+DiME-SALUD2 protocol).
  Arms: Control group (waiting list)
Behavioral: Cognitive Behavioral Treatment (CBT) for smoking cessation — CBT for smoking cessation will be implemented in group-based sessions of four to six patients, once a week over an eight-week period (Becoña, 2007), and includes three different components: (1) Motivational interviewing to stop smoking; (2) Smoking cessation, focused on nicotine fading from the first to the fourth session; (3) Maintenance of abstinence and relapse prevention strategies from the fifth session onwards. This modality of treatment also includes the following components, among others: Therapeutic contract, self-monitoring and graphical representation of tobacco consumption, psychoeducation about tobacco and specific characteristics of smoking behavior, stimulus control, strategies for coping with nicotine withdrawal symptoms, physiological feedback of consumption (using CO and cotinine in urine levels), social reinforcement when meeting nicotine reduction and abstinence goals, training in alternative behaviors to consumption and strategies for the prevention of relapses.
  Arms: Experimental 1: Cognitive-behavioral treatment (CBT) for smoking cessation
Behavioral: CBT for smoking cessation + DiMeSALUD2 protocol — In this group, a training protocol on healthy lifestyle habits and self-management of T2DM will be carried out added to usual care (CBT for smoking cessation). CBT plus DiMe-SALUD2 protocol will be developed as in the precedent group, but with the addition of a psychoeducational protocol for monitoring nicotine fading and abstinence specifically designed to address the particular needs of T2DM smokers. The main components of this protocol will be focused on strengthening healthy lifestyle habits as well as structured around the following core elements: dietary control and healthy nutrition, physical exercise, and glycemic control through daily self-registration of both glycemic variability and nicotine fading or abstinence. If necessary, the therapist will adapt these guidelines according to the established medical advice that the smokers receive from their own endocrinologist, so that this program is developed in accordance with their usual medical care.
  Arms: Experimental 2: CBT for smoking cessation + DiMeSALUD2 protocol

SUMMARY:
The aim of this study is to analyze the effectiveness and efficiency of a multicomponent smoking cessation intervention for Type 2 Diabetes Mellitus (T2DM) smokers, including a training protocol on healthy lifestyle habits and self-management of T2DM called "DiMe-SALUD2" project. Overall, 90 patients will be randomly assigned to one of the following conditions: (1) Control Group (waiting list, n = 30), which will only receive brief psychoeducation advice about smoking cessation; (2) Experimental Group 1 - Cognitive-behavioral treatment (CBT) for smoking cessation (n = 30), where a multicomponent cognitive-behavioral program for quitting will be applied; (3) Experimental Group 2 - CBT for smoking cessation + DiMeSALUD2 protocol (n = 30), where the CBT intervention will be applied plus a training protocol on healthy lifestyle habits and self-management of T2DM.

The specific goals of this project are:

1. To evaluate the added efficacy of the psychoeducation protocol on healthy lifestyle habits and self-management of T2DM plus the multicomponent cognitive-behavioral program to quit smoking (CBT for smoking cessation + DiMeSALUD2 protocol), compared to the standard application of this multicomponent program and to the control group.
2. To describe the impact of the CBT for smoking cessation + DiMeSALUD2 protocol on different key variables (explained below).
3. To analyze the efficiency or cost-effectiveness of the CBT for smoking cessation + DiMeSALUD2 program, and the feasibility of implementing this program in the public health system of Andalusia (Spain).
4. To transfer the knowledge generated to the main health professionals involved in the treatment of smokers with T2DM, through specialized training and the dissemination of a clinical manual created for this purpose.

DETAILED DESCRIPTION:
Despite the fact that there are effective psychological treatments for smoking cessation, studies report that a high percentage of attempts to quit smoking fail and relapse rates after a period of abstinence continue to be high. Thus, it is necessary to incorporate new smoking abstinence and relapse prevention strategies in those treatments implemented with treatment-seeking smokers.

A possible solution to tackle this health problem would be to consider the particular needs of smokers, especially those who have other related pathologies. That is, smoking cessation programs have traditionally been applied to the general population, but there are fewer smoking cessation treatments adapted to the differentiating characteristics of specific groups of the population, especially those who have some type of concurrent physical illness, such as the case of patients with Type 2 Diabetes Mellitus (T2DM). In this sense, smoking behavior is not only related to the etiology of diabetes, but tobacco consumption exerts a harmful effect on these patients, accelerating chronic complications and increasing the risk of mortality.

This study will be conducted through a prospective cohort randomized controlled trial, which will include 90 patients randomly assigned to different conditions:

1. Control Group or waiting list (n = 30), which will only receive brief psychoeducation advice about smoking cessation (that is, participants assigned to this control group will participate in the scheduled assessments but without receiving any of the intensive treatments including in the remaining conditions).
2. Experimental Group 1 - CBT for smoking cessation (n = 30), where a cognitive-behavioral multicomponent program will be implemented in group-based sessions of four to six patients, once a week over an eight-week period.
3. Experimental Group 2 - CBT for smoking cessation + DiMeSALUD2 protocol (n = 30), where the cognitive-behavioral multicomponent program will be applied but adding a specific training protocol on healthy lifestyle habits and self-management of T2DM. The main components of this protocol will be focused on strengthening healthy lifestyle habits and will be structured around the following core elements: dietary control and healthy nutrition, physical exercise, and glycemic control through daily self-registration of both glycemic variability and nicotine fading or abstinence.

On the other hand, the assessment protocol will include their clinical history, different measures of stages of change and nicotine dependence, as well as mental health and quality of life variables. Tobacco consumption will be monitored with biochemical measures (carbon monoxide in exhaled air and cotinine in urine). The efficacy and efficiency of the program will be evaluated at post-treatment and at follow-ups after the end of the intervention (1, 6, and 12 months). This study has been approved by the Ethics Committee of the University of Seville (Ref. 0722-N-22).

The expected results of this research will make it possible to incorporate improvements in routine clinical practice with T2DM smokers, developing a smoking cessation treatment adapted to the specific needs of this population. In addition, this treatment proposal could improve the management of the T2DM disease and comprehensive patient care, as positive impacts are expected that go beyond smoking cessation, such as improved mental health, increased control over possible metabolic changes upon quitting smoking and increased healthy lifestyle habits.

It should be noted that, in the first stage of the DiMe-SALUD2 project, the investigators will conduct a previous pilot study with 15 patients that will be randomly assigned to: 1) Control condition or waiting list; 2) CBT for smoking cessation; 3) CBT for smoking cessation + DiMe-SALUD2 protocol.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18 or over.
* Having smoked 10 or more cigarettes per day within the last year.
* Meeting nicotine dependence criteria (Diagnostic and Statistical Manual of Mental Disorders, fifth Ed.; American Psychiatric Association, 2013).
* Complying with baseline scores equal to or higher than 4 particles per million (ppm) of carbon monoxide (CO) levels in expired air and more than 80 ng/ml of cotinine levels in urine.
* Having a diagnosis of T2DM and receiving routine medical treatment for this condition in their corresponding health services.
* Participants who may present subclinical symptoms of both depression and anxiety will be included.
* Participants who present comorbid physical problems such as cardiorespiratory problems will be included in the study, since smokers with T2DM have a higher incidence of such physical conditions.

Exclusion Criteria:

* Meeting comorbidity with severe psychological or psychiatric disorders, such as bipolar and related disorders, personality disorders, eating disorders (for example, anorexia or bulimia), any disorder included within the schizophrenia spectrum and substance use related disorders (that is, other than nicotine dependence).
* Having a diagnosis of Diabetes Mellitus Type 1 (DMT1) or gestational diabetes.
* Meeting comorbid physical or neurological problems impairing communication. Moreover, we will exclude those patients who do not know the Spanish language enough to hold a fluid conversation.
* Meeting the criteria for any physical health condition whose medical treatment is incompatible or contraindicated for the development of the smoking cessation treatment.
* Receiving other psychological or pharmacological treatment for smoking cessation at the time of recruitment.
* Not being able to attend all treatment sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Smoking abstinence | End of treatment (8-week)
  Includes 24-hours point prevalence abstinence (PPA) (eight weeks). Abstinence will be measured through carbon monoxide (CO) levels (≤ 4 ppm) and cotinine in urine levels (≤ 80 ng/ml).
Smoking abstinence | 1-month follow-up
  Includes 7-day PPA as well as ≤ 4 ppm of carbon monoxide (CO) levels and ≤ 80 ng/ml of cotinine in urine levels.
Smoking abstinence | 6-month follow-up
  Includes 7-day PPA as well as ≤ 4 ppm of carbon monoxide (CO) levels and ≤ 80 ng/ml of cotinine in urine levels.
Smoking abstinence | 12-month follow-up
  Includes 7-day PPA as well as ≤ 4 ppm of carbon monoxide (CO) levels and ≤ 80 ng/ml of cotinine in urine levels.
Mean number of days of smoking continuous abstinence | End of treatment (8-week), 1, 6 and 12 months after treatment completion
  Defined as maintained smoking abstinence since the last time participants smoked, even a puff (since quit day). Abstinence will be measured through carbon monoxide (CO) levels (≤ 4 ppm) and cotinine in urine levels (≤ 80 ng/ml).
Variability of glycemic levels | Pre-treatment, in each treatment sessions (sessions at 1-week, 2-week, 3-week, 4-week, 5-week, 6-week, 7-week), end of treatment (8-week), 1-month, 6-months and 12-months after end of treatment
  Variability of glycemic levels (HbA1c)

SECONDARY OUTCOMES:
Treatment retention | End of treatment (8-week), 1, 6 and 12 months after treatment completion
  Defined as the number of sessions that participants attended during the eight weeks of treatment
Change in the number of cigarettes smoked per day | End of treatment (8-week), 1, 6 and 12 months after treatment completion
  Defined as the reduction in the number of cigarettes smoked per day, since the pre-treatment assessment.
Readiness to change smoking behavior | Pre-treatment, end of treatment (8-week), 1, 6 and 12 months after treatment completion
  Stages of change regarding tobacco use will be evaluated according to the Prochaska and DiClemente's transtheoretical model of change (Prochaska and DiClemente, 1992; Prochaska et al., 1992).
Nicotine dependence | Pre-treatment, end of treatment (8-week), 1, 6 and 12 months after treatment completion
  The Fagerström Test for Nicotine Dependence (Heatherton et al., 1991; Spanish adaptation conducted by Becoña & Vázquez, 1998) will measure changes in nicotine dependence. Total scores range from 0-10, and it includes five levels of dependence (0-2 = very low; 3-4 = low; 5 =moderate; 6-7 = high and 8-10 = very high).
Multidimensional nature of nicotine dependence | Pre-treatment, end of treatment (8-week), 1, 6 and 12 months after treatment completion
  Brief Wisconsin Inventory of Smoking Dependence Motives (Smith et al., 2010) will measure the multidimensional nature of nicotine dependence, including 11 different subscales classified into Primary Dependence Motives (PDM; Automaticity, Craving, Loss of control, and Tolerance) and Secondary Dependence Motives (SDM; Affiliative Attachment, Behavioral Choice/Melioration, Cognitive Enhancement, Cue Exposure/Associative Processes, Negative Reinforcement, Positive Reinforcement, Social/Environmental Goads, Taste/Sensory Properties, and Weight Control). It includes 37 items with a 7-point Likert scale response format. Higher scores indicate higher nicotine dependence (in each subscale).
Anxiety | Pre-treatment, end of treatment (8-week), 1, 6 and 12 months after treatment completion
  State-Trait Anxiety Inventory (Spielberg et al., 1983; Spanish version conducted by Buela-Casal et al., 1982) will assess anxiety symptoms across two subscales: State anxiety and Trait anxiety. Scores in each subscale range from 0-60 (higher percentiles indicate higher state or trait anxiety).
Depressive symptomatology | Pre-treatment, end of treatment (8-week), 1, 6 and 12 months after treatment completion
  Beck's Depression Inventory-Second Edition (Beck et al., 1996; Spanish adaptation of Sanz et al., 2003) will assess the severity of depression. Scores range from 0-63 and it includes different severity levels (0-13 = normal to minimal depression; 20-28 = mild depression; 20-28 = moderate depression; scores above 29 = severe depression).
Diabetes quality of life | Pre-treatment, post-treatment, 1, 6 and 12 months after treatment completion
  Diabetes Quality of Life (Jacobson et al., 1988; Spanish version developed by Reviriego et al., 1996), including four subscales: Satisfaction (rated from 1 very satisfied to 5 very dissatisfied); Impact, Worry (social/vocational) and Worry (DM-related), that are rated from from 1 (no impact/never worried) to 5 (always impacted/ worried). Lower scores indicate higher life satisfaction as well as less impact of diabetes on life.
Diet | Pre-treatment, end of treatment (8-week), 1, 6 and 12 months after treatment completion
  Mediterranean Diet Adherence Screener (MEDAS) (Schröder et al., 2011) will assess adherence to the Spanish Mediterranean diet thought different items regarding the frequency of both food consumption and food habits. We will use the modified version of 13 items recommended by the Andalusian Government and published by Ángel Maqueda et al. (2020), who delete item 8 related to wine consumption. The MEDAS includes dichotomous response options (0 = non-adherent or 1 = adherent to MD) and results equal to or greater than 8 represent good adherence.
Physical activity | Pre-treatment, end of treatment (8-week), 1, 6 and 12 months after treatment completion
  International Physical Activity Questionnaire Short Form (Craig et al., 2003) will collect information on the level of physical activity (high, moderate, low/inactive). It evaluates the minutes of walking during the week, as well as the minutes per week of moderate/vigorous physical activity. Each of the activities assessed must be scored on the basis of METS (Metabolic rate units per minute per week). We will use this short version validated in Spanish by Rodríguez-Muñoz et al. (2017) and recommended by the Andalusian Government (Maqueda et al., 2020; Muñoz et al., 2010].
Anthropometric data | Pre-treatment, end of treatment (8-week), 1, 6 and 12 months after treatment completion
  Body Mass Index
Tobacco Use Disorder Diagnosis | Pre-treatment
  The Structured Clinical Interview for the DSM-5 (SCID-5) (First et al., 2016) will be applied. The SCID-5 evaluates the presence of 11 criteria of nicotine dependence in the last year to establish Tobacco Use Disorder severity (absence, minimal, moderate and severe).

CONTACTS AND LOCATIONS:
Overall Officials: Carla López Núñez, Ph.D, Principal Investigator — Personality, Assessment and Psychological Treatments, School of Psychology, University of Seville
Locations (1):
- Carla López Núñez, Seville, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Nunez C, Fernandez-Artamendi S, Ruiz-Aranda D, Resurreccion DM, Navas-Campana D. A multicomponent smoking cessation program for adults with Type 2 Diabetes Mellitus (DiMe-SALUD2 project): A study protocol of a randomized controlled trial. Contemp Clin Trials Commun. 2024 Aug 28;41:101361. doi: 10.1016/j.conctc.2024.101361. eCollection 2024 Oct. PMID 39290519